CLINICAL TRIAL: NCT03523104
Title: The Chinese Parkinson's Disease With LRRK2 Variants Registry
Brief Title: Chinese PD-LRRK2 Registry
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: CPD-LRRK2R
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — extraction of DNA from peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the Chinese PD-LRRK2 Registry(CPD-LRRK2R) is to develop a database of patients of Parkinson's disease with leucine-rich repeat kinase 2 (LRRK2) gene variants in mainland China.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common disorder among neurodegenerative diseases. LRRK2 missense mutations are the most common known genetic cause of PD. However, some polymorphisms of LRRK2 such as G2385R and R1628P can also affect the risk of developing PD. The investigators aim to establish a database of PD with LRRK2 variants and characterize the clinical manifestation of these patients in mainland China.

Method:

1. Peripheral blood from patients has been tested to have LRRK2 gene variants.
2. Clinical manifestation will be measured by scales and neurological tests. Standard scales include: Unified Parkinson's Disease Rating Scale(UPDRS), Hoehn-Yahr stages, Non-Motor Symptoms Scale (NMSS), mini-mental state examination (MMSE), Parkinson disease sleep scales (PDSS), Rapid Eye Movement Sleep Behaviour Disorder Questionnaire(RBDQ-HK), Epworth Sleepiness Scale (ESS), Rome III functional constipation scale, the Scale for Outcomes in PD for Autonomic Symptoms (SCOPA-AUT), Parkinson Fatigue Scale (PFS), Cambridge-Hopkins Restless Legs Syndrome questionnaire (CHRLSq), Hyposmia rating scale(HRS), Hamilton depression scale, the 39-item Parkinson's Disease Questionnaire(PDQ-39), Freezing of gait scale(FOG), dyskinesia related scales, Wearing-off scale(WO).
3. The investigators will also exam the blood biomarkers of PD such as uric acid and peripheral inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PD by the United Kingdom Parkinson's Disease Society Brain Bank clinical diagnostic criteria or other standard criteria; PD patients detected with positive LRRK2 variants

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PD patients with LRRK2 variants
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Database of Parkinson's disease with LRRK2 variants | 10 years
  Establish the database of Parkinson's disease with LRRK2 variants in mainland China.
Clinical feature | 10 years
  Characterize the clinical feature in patients of Parkinson's disease with LRRK2 variants

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

REFERENCES:
- [Result] Guo JF, Li K, Yu RL, Sun QY, Wang L, Yao LY, Hu YC, Lv ZY, Luo LZ, Shen L, Jiang H, Yan XX, Pan Q, Xia K, Tang BS. Polygenic determinants of Parkinson's disease in a Chinese population. Neurobiol Aging. 2015 Apr;36(4):1765.e1-1765.e6. doi: 10.1016/j.neurobiolaging.2014.12.030. Epub 2015 Jan 6. PMID 25623333
- [Result] Li K, Tang BS, Liu ZH, Kang JF, Zhang Y, Shen L, Li N, Yan XX, Xia K, Guo JF. LRRK2 A419V variant is a risk factor for Parkinson's disease in Asian population. Neurobiol Aging. 2015 Oct;36(10):2908.e11-5. doi: 10.1016/j.neurobiolaging.2015.07.012. Epub 2015 Jul 11. PMID 26234753
- [Result] Yao LY, Guo JF, Wang L, Yu RH, Sun QY, Pan Q, Xia K, Tang BS, Shen L. LRRK2 Pro755Leu variant in ethnic Chinese population with Parkinson's disease. Neurosci Lett. 2011 May 9;495(1):35-8. doi: 10.1016/j.neulet.2011.03.030. Epub 2011 Mar 22. PMID 21406209
- [Result] Wang L, Guo JF, Nie LL, Xu Q, Zuo X, Sun QY, Yan XX, Tang BS. A novel LRRK2 mutation in a mainland Chinese patient with familial Parkinson's disease. Neurosci Lett. 2010 Jan 14;468(3):198-201. doi: 10.1016/j.neulet.2009.10.080. Epub 2009 Oct 29. PMID 19879329
- [Result] Zhang Y, Sun Q, Yi M, Zhou X, Guo J, Xu Q, Tang B, Yan X. Genetic Analysis of LRRK2 R1628P in Parkinson's Disease in Asian Populations. Parkinsons Dis. 2017;2017:8093124. doi: 10.1155/2017/8093124. Epub 2017 Oct 25. PMID 29209554